CLINICAL TRIAL: NCT03967509
Title: Effectiveness of the Cluster Randomized Comet-program Behavioral Preschool Teacher Training in Reducing Externalizing Behavior
Brief Title: Effectiveness of Behavioral Preschool Teacher Training for Externalizing
Acronym: BPTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Social Services Administration (Unknown); Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSA: DNR 3.2-0665/2009; 00-86/2009-36 (Other: National Board of Health and Welfare)
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders; Problem Behavior; Attention Deficit Disorder With Hyperactivity
Keywords: Externalizing behavior problems; Social competence; School readiness; Teacher management training; Cluster randomized effectiveness trial
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Problem Behavior; Attention Deficit Disorder with Hyperactivity; Social Skills | interventions — Comet Assay

STUDY DESIGN:
Intervention Model Description: Preschools randomized to either behavioral teacher training or as waiting list control preschools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral teacher training (Experimental): Behavioral preschool teacher training (BPTT) delivered in an educational group format during nine 2,5-hour biweekly sessions with training at sessions and in between followed by supervisor's feedback on the practice and two optional coaching occasions on the spot.
  Interventions: Behavioral: Comet
- Waiting list control group (No Intervention): Preschool teachers worked with children as usual.

INTERVENTIONS:
Behavioral: Comet
  Other Names: Comet in group format
  Arms: Behavioral teacher training

SUMMARY:
A cluster randomized controlled pre-post effectiveness trial of behavioral preschool teacher training (BPTT) delivered in a practitioner assisted group format for children with externalizing behavior problems. Preschools were randomized to either intervention in 25 preschools or as 22 waiting list control preschools, where teachers in preschool classes with the target child or children were program receivers. Participants were 100 target children 3-5 years old together with 72 enrolled preschool teachers and 83 parents as informants of behavioral outcomes after a five months period of implementation (at six months). The intervention was part of the Swedish evidence-based parent and teacher training programs (Comet) for children and youth with elevated externalizing behavior, and here an adapted version was tried in preschool for the first time. Also investigated was eventual generalized effects to the children's homes and improved social competence as an intermediate mechanism for reduced problem behavior. Effects of implementation fidelity in addition to social acceptability and relevance, such as reliable change, was investigated as well.

DETAILED DESCRIPTION:
Study:

A cluster randomized controlled pre-post effectiveness trial of behavioral preschool teacher training (BPTT) delivered in a practitioner assisted group format for children with externalizing behavior problems. Preschools were randomized to either intervention in 25 preschools or to 22 waiting list control preschools, where preschool classes with the target child or children were program receivers. Informed preschools could apply for participation in the study, then, target children were screened for eligibility. Participants were 100 target children 3-5 years old together with 72 enrolled preschool teachers and 83 parents as informants of behavioral outcomes after a five months period of implementation (at six months).

Intervention:

The intervention was part of the Swedish evidence-based parent and teacher training programs (COmmunication METhod - Comet) for children and youths aged 3-12 and 12-18 years with moderate or elevated externalizing behavior, usually delivered in practitioner assisted group formats but previously evaluated as delivered via internet, single workshops followed by self-administered training, and universal prevention as well. Program implementations and evaluations are executed as collaboration projects between university researchers and the social services administration at place. Intervention content is influenced by operant conditioning, social learning theories, applied behavior analysis, and coercion theory. The focus is to establish a positive and effective interaction and communication style primarily through different reinforcement techniques (e.g., selective attention, more to positive behaviors and less to negative behaviors) and modeling. Parents or teachers meet in psychoeducational group sessions (often 9 to 11 sessions à 2.5 to 3 hours) led by one or two practitioner supervisors. They each follow a comprehensive manual and a highly structured curriculum. Training occurs at sessions (role-plays) and between sessions together with the children, followed-up with feedback in the next session.

Here an adapted version was tried in the preschool setting for the first time. The program corresponded in much to the parent training supplemented with techniques from the school teacher training and a group level administrated glove-puppet play technique to foster children's prosocial skills. (Results from the universal part of the program are not reported.) The nine sessions curriculum consisted of 2.5-hour biweekly meetings and two optional visits from supervisors with coaching on the spot. Practitioner supervisors (n = 27) were educated by a cognitive-behavior oriented psychologist during five days term one and two days term two.

Investigation issues:

The primary aim was to investigate behavioral outcome effects of the preschool teacher program. Would effects (Cohen's d) be in the medium-large range as found for Comet parent training (i.e., d = .50-.90) or in the small-medium range as often found for preventive developmental preschool programs (i.e., d = .20-.40)? With effects of about .40, a sample size restricted to 100 subjects, and an alpha at .05, power would be close to sufficient (i.e., .70). Of interest was to compare the effects of this program with effects found for other preschool program investigations of externalizing behavior problems.

Also investigated was eventual generalized effects to the children's homes. Of what magnitude would such effects be, if any, and would the parents' ratings validate the teachers' ratings, and thus, support the intervention? Such effects may have implications for future implementations, for example if the program is sufficiently efficient as a stand-alone intervention in reducing externalizing behavior problems or not sufficiently efficient. There was also a question of degree of informants agreement/discrepancy. Furthermore, would improved prosocial and regulatory skills function as a predictive and an intermediate mechanism for reduced problem behavior, and/or would there be room for other intervention features to contribute as well? In addition, as a trial in the real world, effects of implementation fidelity as well as social acceptability and relevance, such as proportions of children with reliable change, were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Elevated level of externalizing behavior
* Exceeding cutoff value 11 on the Strengths and Difficulties Questionnaire, total scale

Exclusion Criteria:

-

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-08-18 (Actual); Primary Completion 2011-02-03 (Actual); Study Completion 2011-02-03 (Actual)

PRIMARY OUTCOMES:
Sutter-Eyberg Student Behavior Inventory (SESBI) | Change measures: baseline (pre) and after 6 months (post).
  A rating scale for teachers measuring child externalizing behaviors. The two subscales Intensity (range 38-266) representing frequency, severity, or level of problem behaviors occurring from never (1) to always (7) and Problem (range 0-38) reflecting behaviors that are perceived as problems or not are reported independently. Higher values indicate more externalizing behaviors or more problems.
Eyberg Child Behavior Inventory (ECBI) | Change measures: baseline (pre) and after 6 months (post).
  A rating scale for parents measuring child externalizing behaviors. The two subscales Intensity (range 36-252) representing frequency, severity, or level of problem behaviors occurring from never (1) to always (7) and Problem (range 0-36) reflecting behaviors that are perceived as problems or not are reported independently. Higher values indicate more externalizing behaviors or more problems.
Social Competence Scale (SCS) | Change measures: baseline (pre) and after 6 months (post).
  A rating scale for teachers and parents estimating child prosocial behavior, communicative skills, and self-control containing two 5-point subscales with six items each; Prosocial (e.g., solve conflicts, share, helpful, listen, not bossy) and Emotional regulation (e.g., can accept a failure, calm down, think before acting, control temper). The total score may vary between 12 and 60. Higher values indicate better social competence.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) Supplement - Impact and Burden | Change measures: baseline (pre) and after 6 months (post).
  A rating scale for teachers and parents asking about child difficulties with emotions, concentration, behavior, and getting on with other people on a 4-point scale from no difficulties to severe difficulties. Consecutive items (three for teachers and five for parents) ask about child distress and social impairment in the domains of home life, friendships, classroom learning, and leisure activities. Total range for teachers was 0-12 (first question included) and total range for parents was 0-15 (first question excluded). Last, a burden item asks if the difficulties put a burden on the family or the preschool from not at all to much (range 0-3). Impact and Burden are reported separately. Higher values indicate more negative impact and burden because of behavior problems.

OTHER OUTCOMES:
Credibility/Expectancy Questionnaire | At baseline (pre).
  Teachers and supervisors rated how much they believed in the method and their expectations of improvement in terms of five items covering reasonableness, degree of belief in magnitude of impact on externalizing and other behavior problems, willingness to recommend, and expectation of improvement of the preschool situation on a 10-point scale from not at all to much. Total mean score could vary between 1 and 10, where higher score means higher credibility/expectancy beliefs.
Program fidelity, teacher | Reported per 9 biweekly sessions after intervention at 5 months.
  Teachers reported on program fidelity per session: attendance and number of program components/techniques accomplished. Session attendance was reported as the ratio of attending teachers to participating teachers for each session. Accomplishment and techniques used were categorized as educational themes (0-1, max = 36), role-plays (0-2: none, observing other roleplay, own role-play, max = 22), homework assignments (0-1 or 2, max = 33), and feedback on training between sessions (0-2: none, some, detailed, max = 16). Teacher fidelity measures were reported as means per program component and percentage of accomplishment.
Program fidelity and teacher reliability check, supervisor | After intervention at 5 months.
  Supervisors reported on four fidelity themes: 1. Self-report on manual content completed. 2. Three ratings of teacher accomplishment: 2. session attendance, 3. role-plays, and 4. homework assignments completed on a 5-point scale from not at all to fully. Supervisor fidelity measure was reported as total mean and percentage of accomplishment.
Consumer satisfaction, teacher | After intervention at 5 months.
  Preschool teachers rated perceived 1. effectiveness, 2. comprehension of the methods, and 3. support of their professional role on a 4-point scale from not at all (1), little (2), pretty much (3), to very (4). Reported as percentage of teachers per category.
Consumer satisfaction, supervisor | After intervention at 5 months.
  Supervisors reported on support and time for their work from their employer on a 4-point categorical scale from neither support or time (1), time, but lack of support (2), support, but lack of time (3) to both support and time (4) reported in percentages per category.
Motivation | After intervention at 5 months.
  Motivation to participate in the program was rated by teachers and supervisors on 4 scale steps from not at all to very motivated and reported in percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Åsa K Kling, PhD student, Principal Investigator — Uppsala University; Mats Fredrikson, Professor, Study Chair — Uppsala University
Locations (1):
- Komet [Comet] Programs, Stockholm, Johanneshov, Sweden

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, CSR
Time Frame: Three months after publication and five years hereafter.
Access Criteria: If similar type of data including measures (all IPD) are available elsewhere, and it is possible to aggregate data, then a data collaboration project might be a possibility.

REFERENCES:
- [Background] Eyberg, S., Pincus, D. Eyberg Child behavior Inventory (ECBI) and Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R). Professional manual. Odessa, Florida: PAR, 1999.
- [Background] Conduct Problems Prevention Research Group. Social Competence Scale (Parent), 1995. Retrieved from the Fast Track Project: http://www.fasttrackproject.org
- [Result] Kling A, Forster M, Sundell K, Melin L. A randomized controlled effectiveness trial of parent management training with varying degrees of therapist support. Behav Ther. 2010 Dec;41(4):530-42. doi: 10.1016/j.beth.2010.02.004. Epub 2010 Oct 1. PMID 21035616
- [Result] Enebrink P, Hogstrom J, Forster M, Ghaderi A. Internet-based parent management training: a randomized controlled study. Behav Res Ther. 2012 Apr;50(4):240-9. doi: 10.1016/j.brat.2012.01.006. Epub 2012 Jan 30. PMID 22398153
- [Result] Forster, M., Sundell, K., Morris, R, Karlberg, M., Melin, L. A randomized controlled trial of a standardized behavior management intervention for students with externalizing behavior. Journal of Emotional and Behavioral Disorders, 20(3): 169-183, 2012
- [Result] Forster, M., Kling, Å., Sundell, K. Clinical significance of parent training for children with conduct problems. International Journal of Conflict and Violence, 6(2): 187-200, 2012.
- [Result] Ghaderi A, Kadesjo C, Bjornsdotter A, Enebrink P. Randomized effectiveness Trial of the Family Check-Up versus Internet-delivered Parent Training (iComet) for Families of Children with Conduct Problems. Sci Rep. 2018 Jul 31;8(1):11486. doi: 10.1038/s41598-018-29550-z. PMID 30065246
- [Result] Hogstrom J, Olofsson V, Ozdemir M, Enebrink P, Stattin H. Two-Year Findings from a National Effectiveness Trial: Effectiveness of Behavioral and Non-Behavioral Parenting Programs. J Abnorm Child Psychol. 2017 Apr;45(3):527-542. doi: 10.1007/s10802-016-0178-0. PMID 27334706
- [Result] Stattin H, Enebrink P, Ozdemir M, Giannotta F. A national evaluation of parenting programs in Sweden: The short-term effects using an RCT effectiveness design. J Consult Clin Psychol. 2015 Dec;83(6):1069-1084. doi: 10.1037/a0039328. Epub 2015 May 25. PMID 26009784
- [Result] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Result] Goodman R. The extended version of the Strengths and Difficulties Questionnaire as a guide to child psychiatric caseness and consequent burden. J Child Psychol Psychiatry. 1999 Jul;40(5):791-9. PMID 10433412
- [Result] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Result] Malmberg M, Rydell AM, Smedje H. Validity of the Swedish version of the Strengths and Difficulties Questionnaire (SDQ-Swe). Nord J Psychiatry. 2003;57(5):357-63. doi: 10.1080/08039480310002697. PMID 14522609
- [Result] Axberg U, Johansson Hanse J, Broberg AG. Parents' description of conduct problems in their children - a test of the Eyberg Child Behavior Inventory (ECBI) in a Swedish sample aged 3-10. Scand J Psychol. 2008 Dec;49(6):497-505. doi: 10.1111/j.1467-9450.2008.00670.x. Epub 2008 Aug 12. PMID 18705675
- [Result] Conduct Problems Prevention Research Group. Social Competence Scale (Parent) - Technical reports, 1995-2002. Retrieved from: http://www.fasttrackproject.org